CLINICAL TRIAL: NCT05838820
Title: Reliability of the Jebsen-Taylor Hand Function Test and the Nine-Hole Peg Test in Individuals With Carpal Tunnel Syndrome: A Cross-sectional Study
Brief Title: Hand Function Tests in Carpal Tunnel Syndrome: A Cross-sectional Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Lecturer of Physical Therapy and Director of Electromyography Lab, Ahram Canadian University
Other Study IDs: 012/005988
Record Dates: First submitted 2023-04-19; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Carpal Tunnel Syndrome (CTS) Group: This group will consist of individuals diagnosed with carpal tunnel syndrome (CTS) who are 18 years of age or older and who are able to provide informed consent to participate in the study. The group will be recruited from a single center and will be asked to complete the Jebsen-Taylor Hand Function Test and the Nine-Hole Peg Test twice, with a 1-week interval between the two assessments. The aim is to establish the test-retest reliability of these tests in individuals with CTS. The group will include at least 50 participants and will be diverse in terms of age, gender, and race/ethnicity to ensure that the study findings are generalizable to a broader population.
  Interventions: Diagnostic Test: Nine-Hole Peg Test; Diagnostic Test: Jebsen-Taylor Hand Function Test

INTERVENTIONS:
Diagnostic Test: Nine-Hole Peg Test — The Nine-Hole Peg Test is a standardized test that measures manual dexterity and finger movement speed in individuals with hand impairments. The test involves the placement of nine pegs in a pegboard, one at a time, and then removal of each peg as quickly as possible using one hand. The test is timed, and the time required to complete the test provides an indication of manual dexterity and finger movement speed. The Nine-Hole Peg Test has been previously validated and is commonly used in clinical practice.
Diagnostic Test: Jebsen-Taylor Hand Function Test — is a standardized test that assesses fine motor skills and functional abilities of the hand. The test involves the completion of seven subtests, including writing, simulated page turning, picking up small objects, stacking checkers, lifting large objects, simulated feeding, and stacking cans. Each subtest is timed, and the time required to complete each subtest provides an indication of hand function. The Jebsen-Taylor Hand Function Test has been previously validated and is commonly used in clinical practice.

SUMMARY:
This is a cross-sectional study that aims to establish the test-retest reliability of two standardized tests (Jebsen-Taylor Hand Function Test and Nine-Hole Peg Test) in individuals with carpal tunnel syndrome (CTS). The study will involve at least 50 participants with CTS who will complete the tests twice, with a 1-week interval between the two assessments. The test-retest reliability will be assessed using intraclass correlation coefficient (ICC) and Bland-Altman plots. The study is expected to provide information on the reliability of these tests in individuals with CTS, which can help clinicians more accurately assess hand function and monitor treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with carpal tunnel syndrome (CTS)
* 18 years of age to 60 years old
* Able to provide informed consent to participate in the study

Exclusion Criteria:

* History of hand or wrist surgery within the past 6 months
* Severe hand or wrist pain that would prevent completion of the tests
* Severe cognitive impairment or language barrier that would prevent understanding of the test instructions
* Any other medical condition that could affect hand function or interfere with test completion
* Participation in any other clinical trial or research study involving the hand or wrist within the past 3 months
* Inability to comply with study procedures or follow-up requirements

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population will consist of individuals diagnosed with carpal tunnel syndrome (CTS) who are 18 years of age or older and who are able to provide informed consent to participate in the study. Participants will be recruited from a single center and will be diverse in terms of age, gender, and race/ethnicity to ensure that the study findings are generalizable to a broader population.
  Participants will be excluded from the study if they have a history of hand or wrist surgery within the past 6 months, severe hand or wrist pain that would prevent completion of the tests, severe cognitive impairment or language barrier that would prevent understanding of the test instructions, any other medical condition that could affect hand function or interfere with test completion, participation in any other clinical trial or research study involving the hand or wrist within the past 3 months, or inability to comply with study procedures or follow-up requirements.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-05-18 (Estimated); Primary Completion 2023-09-27 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Test-Retest Reliability of Jebsen-Taylor Hand Function Test and Nine-Hole Peg Test in Individuals with Carpal Tunnel Syndrome | 1-week interval between the two assessments
  The primary outcome measure of this study is the test-retest reliability of the Jebsen-Taylor Hand Function Test and the Nine-Hole Peg Test in individuals with carpal tunnel syndrome (CTS). Test-retest reliability will be assessed using the intraclass correlation coefficient (ICC) and Bland-Altman plots.

SECONDARY OUTCOMES:
Correlation with clinical measures | 1-week interval between the two assessments
  This secondary outcome measure assesses the inter-rater reliability of the Jebsen-Taylor Hand Function Test and the Nine-Hole Peg Test in individuals with carpal tunnel syndrome (CTS). This will involve comparing the results of the tests administered by two different raters to determine the consistency of the results.

CONTACTS AND LOCATIONS:
Overall Officials: Amal Fawzy, Ph.d, Study Chair — Faculty of Physical Therapy, Ahram Canadian University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD) collected during this study will be available upon reasonable request. Requests for access to the data should be submitted via email to mohamed.elmeligie@acu.edu.eg. All requests will be reviewed by the study investigators to ensure that they are reasonable and consistent with the ethical principles of the study. Access to the data will be granted in compliance with applicable laws and regulations, and with appropriate safeguards to protect the privacy and confidentiality of study participants.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After the trial ends and up to 1 year post trial.
Access Criteria: via email to mohamed.elmeligie@acu.edu.eg